CLINICAL TRIAL: NCT01067300
Title: A Prospective, Multicenter Randomized Study Comparing Single Versus Double Umbilical Cord Blood Transplantation in Children and Young Adults (<35 Years) With Acute Leukemia Remission
Brief Title: A Study Comparing Single Versus Double Umbilical Cord Blood Transplantation in the Young With Acute Leukemia Remission
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2009-17; 2009-A00792-55
Record Dates: First submitted 2010-02-10; First posted 2010-02-11 (Estimated); Last update posted 2015-10-01 (Estimated); Status verified 2015-09

CONDITIONS: Leukemia
Keywords: young; acute leukemia in remission; Children or young adults (< 35 years) with acute leukemia in remission
MeSH Terms: conditions — Leukemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Double unit unrelated cord blood transplantation (Active Comparator): Transplantation of unrelated cord blood units is done at least 24 hours after last chemotherapy and carried out during the same day. The unit presenting the best degree of HLA compatibility with the patient will be transfused in first. If the 2 units have the same degree of HLA compatibility with the recipient, the unit with the higher cell dose will be transfused in first. A 2 hours time interval between the 2 transfusions will be respected.
  Interventions: Procedure: Transplantation of unrelated cord blood unit(s)
- single unit unrelated cord blood transplantation (Active Comparator): Transplantation of a single unrelated cord blood unit at least 24 hours after last chemotherapy
  Interventions: Procedure: Transplantation of unrelated cord blood unit(s)

INTERVENTIONS:
Procedure: Transplantation of unrelated cord blood unit(s) — Myeloablative conditioning regimen includes, according to the patient age, either total body irradiation, fludarabine and cyclophosphamide with a GvHD prophylaxis based on cyclosporine A and mycophenolate, or the association busulfan, cyclophosphamide and anti-thymocyte globulin with GvHD prophylaxis being cyclosporine A and steroids.
  Other Names: Infusion of unrelated cord blood unit(s)

SUMMARY:
Unrelated cord blood transplantation (UCBT) has been used for several years when there is no HLA identical sibling or unrelated donor.Since the recent publication of encouraging results after transplantation of two UCB units, the number of these double-transplantations increases in a very significant way.However, there is currently no prospective study comparing in a reliable way the double-transplantation to single-transplantation results.The investigators propose a prospective and randomized study comparing the results of single versus double unit UCBT in children and young adults (< 35 yrs) with acute leukemia in remission. This is an open, multicenter study carried out in the allogeneic transplant centers from the French society for hematopoietic stem cell transplantation and cell therapy. The primary objective is to compare the incidence of transplantation failure in the two treatment arms. Transplantation failure, the primary endpoint of the study, is defined by the occurrence of one of the following events : transplant-related death, second allogeneic transplantation or autologous backup infusion for primary engraftment failure, autologous recovery. The financial impact of these double-transplantations being to date unknown, the project also includes a cost-effectiveness study, the effectiveness criterion being a decrease in transplantation failure incidence. The secondary clinical endpoints are: overall survival and disease-free survival, relapse incidence, transplant-related mortality, incidence of severe infections and GvHD. The secondary biological endpoints are: hematological and immunological recovery, post transplant chimerism.

DETAILED DESCRIPTION:
Background and rationale:

Unrelated cord blood transplantation (UCBT) has been used for several years when there is no HLA identical sibling or unrelated donor. During the year 2007, 218 of the 783 unrelated hematopoietic stem cell transplantation (28%) carried out in France were UCBT. This proportion is 37% in children (58/157). Clinical outcome after UCBT strongly depends on the transplant cell dose. Since the recent publication of encouraging results after transplantation of two UCB units, the number of these double-transplantations increases in a very significant way. Thus 121/218 UCBT performed in France during 2007 were double-transplantations (55%) whereas this proportion was 81/180 (45%) in 2006, 30/144 (21%) in 2005, 5/77 (6%) in 2004 and 0/44 in 2003. However, there is currently no prospective study comparing in a reliable way the double-transplantation to single-transplantation results.

Study design:

The investigators propose a prospective and randomized study comparing the results of single versus double unit UCBT in children and young adults (< 35 yrs) with acute leukemia in remission. This is an open, multicenter study carried out in the allogeneic transplant centers from the French society for hematopoietic stem cell transplantation and cell therapy (Société Française de Greffe de Moelle et de Thérapie Cellulaire, SFGM-TC).

Objectives:

The primary objective is to compare the incidence of transplantation failure in the two treatment arms. Transplantation failure, the primary endpoint of the study, is defined by the occurrence of one of the following events : transplant-related death, second allogeneic transplantation or autologous backup infusion for primary engraftment failure, autologous recovery. The financial impact of these double-transplantations being to date unknown, the project also includes a cost-effectiveness study, the effectiveness criterion being a decrease in transplantation failure incidence. The secondary clinical endpoints are: overall survival and disease-free survival, relapse incidence, transplant-related mortality, incidence of severe infections and GvHD. The secondary biological endpoints are: hematological and immunological recovery, post transplant chimerism.

Methods:

Transplantation methods: Myeloablative conditioning regimen includes, according to the patient age, either total body irradiation, fludarabine and cyclophosphamide with a GvHD prophylaxis based on cyclosporine A and mycophenolate, or the association busulfan, cyclophosphamide and anti-thymocyte globulin with GvHD prophylaxis being cyclosporine A and steroids.

Statistical methods: The experimental schedule is based on a multiple testing procedure, using the method described by O' Brien and Fleming. This offers the possibility of stopping the trial before the end of inclusions if a significant difference between the two arms occurs. In this trial, two sequential analyses are planned: an interim analysis at 18 months and a final analysis at 36 months. Probabilities of survival and DFS are estimated according to the Kaplan-Meier method. In the presence of one or several competitive risks, the cumulative incidence of an event is estimated according to the method of Gray. Thus, relapse is a competing risk for transplantation failure in the study primary endpoint evaluation. Comparisons between the two treatment arms are carried out by the Log rank test for Kaplan-Meier estimates and by the Gray's test for the cumulated incidences. The intent to treat analysis (according to the random allocation) will be preferred to a per-protocol analysis which will be an additional analysis. An independent committee will be made up in order to control the decisions of study continuation or stopping at time of the interim analysis.

Sample calculation, study feasibility and duration:

In the setting of a sequential trial including one interim analysis, with a cumulated incidence of transplantation failure hypothesis being 40% in the single-transplantation and 20% in the double-transplantation arm (alpha risk, 5%, power, 80%, 5% non evaluable patients), the estimate of sample size is 99 by group, i.e. a total of 198. Taking into account the UCBT activity in France (data from the French biomedicine agency), the enrolment phase of the study is planned to last 30 months. Minimum post-transplant follow-up duration being 6 months, duration of the study is 3 years.

ELIGIBILITY:
Inclusion Criteria:

* age < 35 years
* acute leukemia in remission which need unrelated transplantation
* lack of a suitable unrelated donor
* availability of at least 2 UCB units 4/6, 5.6 or 6/6 HLA identical to the patient and between them, which contain more than 3 x 107 nucleated cells per kilogram of recipient for the first unit and more than de 1.5 x 107 nucleated cells per kilogram of recipient for the second
* general status compatible with a myéloablative conditioning regimen

Exclusion Criteria:

* availability of an HLA identical sibling
* availability of an unrelated donor considered to be acceptable by the transplant center
* History of allogeneic stem cell transplantation
* History of a total body irradiation
* Organ failure or patient general status considered to be incompatible with a myeloablative conditioning regimen
* Active psychiatric disease
* Uncontrolled bacterial, viral or fungal infection
* Positive HIV serology
* Pregnancy

Max Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 198 (Estimated)
Dates: Start 2010-02; Primary Completion 2016-01 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
to compare the incidence of transplantation failure in the two treatment arms. | 3 years

SECONDARY OUTCOMES:
a cost-effectiveness study, the effectiveness criterion being a decrease in transplantation failure incidence. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Gerard MICHEL, Principal Investigator — Assistance Publique - Hôpitaux de Marseille
Locations (1):
- Assistance Publique - Hôpitaux de Marseille, Marseille, France

REFERENCES:
- [Derived] Michel G, Galambrun C, Sirvent A, Pochon C, Bruno B, Jubert C, Loundou A, Yakoub-Agha I, Milpied N, Lutz P, Marie-Cardine A, Gandemer V, Blaise D, Michallet M, Rialland F, Renard C, Oudin C, Esmiol S, Seux M, Baumstarck K, Mohty M, Rocha V, Dalle JH. Single- vs double-unit cord blood transplantation for children and young adults with acute leukemia or myelodysplastic syndrome. Blood. 2016 Jun 30;127(26):3450-7. doi: 10.1182/blood-2016-01-694349. Epub 2016 Apr 20. PMID 27099151